CLINICAL TRIAL: NCT05714696
Title: Mechanisms Explaining the Link Between Weight Discrimination and Poor Cardiovascular Health
Brief Title: Weight Discrimination and Poor Cardiovascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mary Gerend, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: R56HL159177 (NIH); R56HL159177 (NIH)
Record Dates: First submitted 2023-01-06; First posted 2023-02-06 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight discrimination experience (Experimental): Participants in the experimental condition will:
  1. Learn that their group mates are biased against overweight people (i.e., they have negative attitudes toward people with higher body weight),
  2. Receive feedback about their personal attributes that is consistent with negative weight-based stereotypes (e.g., lacking self-discipline), and
  3. Not be selected as a partner for the remaining lab tasks (i.e., this experience may prompt feelings of social exclusion).
  Interventions: Behavioral: Weight discrimination experience
- Control experience (Active Comparator): Participants in the control condition will:
  1. Learn that their group mates are very accepting of overweight people (i.e., they have positive attitudes toward people with higher body weight),
  2. Receive positive feedback about their personal attributes that is not consistent with negative weight-based stereotypes, and
  3. Will be told that one of their group members had to leave early for an emergency so the pairs cannot be assembled as usual (i.e., this experience should not prompt feelings of social exclusion).
  Interventions: Behavioral: Control experience

INTERVENTIONS:
Behavioral: Weight discrimination experience — In the experimental condition, participants will learn that their group members are biased against overweight people but not elderly or racial/ethnic minority individuals, as indicated by the "getting to know you" summary ratings handout. Participants will also receive negative feedback about their personal attributes by being labeled with negative weight-based stereotypes. Although some ratings will be positive (e.g., they will receive high ratings on being friendly and kind), participants will be rated poorly on attributes viewed as necessary to develop a strong marketing campaign (i.e., motivation to work hard, possessing self-discipline to persist at the task, and competence). After (ostensibly) assembling the group's preferences, the experimenter will inform participants that no one selected them to be their partner, thus they will perform the next few tasks alone. This manipulation has been shown to prompt feelings of social exclusion.
  Arms: Weight discrimination experience
Behavioral: Control experience — In the control condition, participants will learn that their group members have positive attitudes toward people with higher body weight, as well as elderly and racial/ethnic minority individuals, as indicated by the "getting to know you" summary ratings handout. Participants will also receive positive feedback about their personal attributes, as indicated by the summary ratings averaged across the three members. Finally, participants in the control condition will be told that one of their group members had to leave unexpectedly for a family emergency, so pairs cannot be assembled as usual, thus they will perform the next few tasks alone. This manipulation should not prompt feelings of social exclusion.
  Arms: Control experience

SUMMARY:
People with obesity regularly experience discrimination on the basis of their body weight and such experiences are associated with increased risk for poor cardiovascular health. The goal of this clinical trial is to identify cognitive, affective, behavioral, and physiological factors that explain the relationship between weight discrimination and poor health outcomes.

A diverse sample of adults with obesity will be randomly assigned to a social interaction encounter that simulates a typical weight discrimination experience (experimental manipulation) vs. a control manipulation that does not involve discrimination. The investigators will examine the immediate effects of the experimental manipulation on cognitive (e.g., self-regulation), affective (e.g., negative emotion), behavioral (e.g., comfort eating), and physiological (e.g., cortisol secretion) outcomes.

Two additional aims of the study are to identify psychological traits that moderate responses to weight discrimination and to assess whether the negative health effects of weight discrimination differ by age, sex/gender, race, or ethnicity.

DETAILED DESCRIPTION:
Discrimination is a critical social determinant of health that underlies poor health outcomes. One common but understudied form of discrimination is weight discrimination. Weight discrimination is the behavioral manifestation of weight stigma-the social devaluation of people with excess body weight. Findings suggest that the stress produced by weight discrimination prompts weight gain, creating a vicious cycle between weight discrimination and obesity. Further, there is now well-documented evidence that experiencing weight discrimination is associated with increased risk for cardiovascular disease. Little is known, however, about mechanisms explaining the link between weight discrimination and poor cardiovascular health. Using a rigorous experimental approach, this project will identify mechanisms through which weight discrimination harms health. Findings will facilitate the long-term goal of this research: interventions to decrease the negative health consequences of weight discrimination.

As a step toward this goal, this project proposes to conduct an experiment in which a diverse sample of adults with obesity will be randomly assigned to experience (vs. not experience) weight discrimination in a controlled experimental setting. Drawing on previous research and the investigators' pilot data, the interpersonal context chosen for the study simulates situations in which people with obesity commonly experience weight discrimination in their daily lives (e.g., employment settings).

The study will involve two parts: a pre-session baseline survey and an experimental session that will take place in the lab. The baseline survey will be completed online and will assess individual difference variables/psychological variables and demographic characteristics. The in-person lab visit will take place on campus about one week after completion of the baseline survey. The study manipulation (i.e., intervention) will be delivered during the lab visit. Primary outcome variables will be assessed during the lab visit, after delivery of the intervention.

The following aims will be tested: (1) Identify early-stage cognitive, affective, behavioral, and physiological mechanisms activated by experimentally manipulated weight discrimination; (2) Identify psychological variables (e.g., internalized weight bias) that moderate effects of weight discrimination; and (3) Identify demographic characteristics (e.g., gender, race) that moderate effects of weight discrimination. Exposure to weight discrimination (vs. control) is hypothesized to result in elevated responses on early-stage mechanisms that culminate in poor cardiovascular health (e.g., impaired self-regulation, higher negative emotion, more social withdrawal and comfort eating, increased cortisol secretion). This research will identify novel and highly modifiable targets for interventions designed to reduce the negative health effects of weight discrimination. In testing moderator variables, this work will identify individuals who display vulnerability vs. resilience to the harmful effects of discrimination. Information about moderators will thus help future intervention efforts target those individuals most likely to benefit from intervention. Given the high prevalence of obesity and the millions of Americans affected by weight discrimination, this research will address a crucial public health issue.

ELIGIBILITY:
Inclusion Criteria:

* (1) body mass index (BMI) greater than or equal to 30 (units: weight in kilograms divided by height in meters squared; BMI criteria for obesity)
* (2) 18 years of age or older
* (3) able to read and understand English
* (4) have Internet access (to complete the baseline survey)
* (5) able to come to FSU's campus to take part in a lab-based study

Exclusion Criteria:

* (1) having participated in any of our pilot studies on weight stigma
* (2) diagnosed with a current major psychiatric disorder (e.g., major depressive disorder, eating disorder)
* (3) pregnant or nursing
* (4) diagnosed with Cushing syndrome or taking steroid-based medications
* (5) having allergies to ingredients in the foods being offered during the taste test (e.g., gluten, peanuts).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2023-02-05 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary A Gerend, PhD, Principal Investigator — Florida State University, College of Medicine
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team agrees to develop a transportable de-identified database, codebook, and mechanism by which data could be shared with other investigators upon approval of the PI.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available 9 months after completion of the trial and will be made accessible up to 36 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial data can be requested by qualified researchers engaging in independent scientific research. Investigators will be asked to complete a standardized request form stating the specific aims of the analysis, the analytic plan, resources the requestors have to carry out the project, the proposed timeline, and distribution goals (manuscripts and/or grant application). The PI will review these requests to determine whether the proposed analyses constitute an innovative and significant exploration of the data, whether the proposed team has sufficient resources to undertake the request, how data will be protected/managed, and whether there are sufficient resources to honor the request. If any of these issues are problematic, the PI will attempt to negotiate a fair resolution with the interested parties and/or with NIH program staff. The PI will keep a record of all individuals/research teams who receive a copy of the data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the local community between February 2023 and April 2024. The first participant was enrolled on February 5, 2023 and the last participant was enrolled on April 26, 2024.
Pre-assignment Details: Of 333 enrolled participants, 271 were randomized to experimental condition.
Groups:
- Weight Discrimination Experience: Participants in the experimental condition will:
  1. Learn that their group mates are biased against overweight people (i.e., they have negative attitudes toward people with higher body weight),
  2. Receive feedback about their personal attributes that is consistent with negative weight-based stereotypes (e.g., lacking self-discipline), and
  3. Not be selected as a partner for the remaining lab tasks (i.e., this experience may prompt feelings of social exclusion).
  Weight discrimination experience: In the experimental condition, participants will learn that their group members are biased against overweight people but not elderly or racial/ethnic minority individuals, as indicated by the "getting to know you" summary ratings handout. Participants will also receive negative feedback about their personal attributes by being labeled with negative weight-based stereotypes. Although some ratings will be positive (e.g., they will receive high ratings on being friendly and kind), participants will be rated poorly on attributes viewed as necessary to develop a strong marketing campaign (i.e., motivation to work hard, possessing self-discipline to persist at the task, and competence). After (ostensibly) assembling the group's preferences, the experimenter will inform participants that no one selected them to be their partner, thus they will perform the next few tasks alone. This manipulation has been shown to prompt feelings of social exclusion.
- Control Experience: Participants in the control condition will:
  1. Learn that their group mates are very accepting of overweight people (i.e., they have positive attitudes toward people with higher body weight),
  2. Receive positive feedback about their personal attributes that is not consistent with negative weight-based stereotypes, and
  3. Will be told that one of their group members had to leave early for an emergency so the pairs cannot be assembled as usual (i.e., this experience should not prompt feelings of social exclusion).
  Control experience: In the control condition, participants will learn that their group members have positive attitudes toward people with higher body weight, as well as elderly and racial/ethnic minority individuals, as indicated by the "getting to know you" summary ratings handout. Participants will also receive positive feedback about their personal attributes, as indicated by the summary ratings averaged across the three members. Finally, participants in the control condition will be told that one of their group members had to leave unexpectedly for a family emergency, so pairs cannot be assembled as usual, thus they will perform the next few tasks alone. This manipulation should not prompt feelings of social exclusion.
Period: Overall Study
Arm/Group | Weight Discrimination Experience | Control Experience
Started | 136 | 135
Completed | 136 | 135
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Weight Discrimination Experience | Control Experience | Total
Number analyzed (Participants) | 136 | 135 | 271
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.99 (13.41) | 38.70 (13.28) | 38.34 (13.33)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 109 | 108 | 217
  Male | 26 | 26 | 52
  Prefer not to answer | 0 | 1 | 1
  Unknown | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 16 | 32
  Not Hispanic or Latino | 120 | 119 | 239
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 43 | 41 | 84
  White | 77 | 85 | 162
  More than one race | 5 | 5 | 10
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 136 | 135 | 271
Body mass index [Mean (Standard Deviation); unit: kg/m2] — Body mass index was derived from participants' measured height and weight and is reported in kg/m2.
  kg/m2 | 37.99 (6.99) | 37.22 (5.73) | 37.61 (6.39)

OUTCOME MEASURES:

1. Primary Outcome: Negative Affect
Description: A modified version of the Positive and Negative Affect Scale-Expanded Form (PANAS-X) will be used to assess emotions in response to the experimental manipulation. The scale demonstrates good validity and reliability. Emotions will be assessed with 46 adjectives (e.g., angry, confident) by indicating the extent to each emotion is felt at that moment (1=very slightly or not at all to 5=extremely). A composite score for negative affect will be created by taking the average of the relevant adjectives. Scores will range from 1 to 5, with higher scores indicating more negative emotion.
Time Frame: 2 minutes after delivery of the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Weight Discrimination Experience | Control Experience
Number analyzed (Participants) | 136 | 135
score on a scale | 1.43 (0.49) | 1.29 (0.33)
Statistical Analysis 1: Comparison: Control Experience; Test type: Superiority; p = .007, t-test, 2 sided

2. Primary Outcome: Positive Affect
Description: A modified version of the Positive and Negative Affect Scale-Expanded Form (PANAS-X) will be used to assess emotions in response to the experimental manipulation. The scale demonstrates good validity and reliability. Emotions will be assessed with 46 adjectives (e.g., angry, confident) by indicating the extent to each emotion is felt at that moment (1=very slightly or not at all to 5=extremely). A composite score for positive affect will be created by taking the average of the relevant adjectives. Scores will range from 1 to 5, with higher scores indicating more positive emotion.
Time Frame: 2 minutes after delivery of the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Weight Discrimination Experience | Control Experience
Number analyzed (Participants) | 136 | 135
score on a scale | 2.83 (0.94) | 3.04 (0.82)
Statistical Analysis 1: Comparison: Control Experience; Test type: Superiority; p = .049, t-test, 2 sided

3. Primary Outcome: Self-efficacy for Weight Control Behavior
Description: Self-efficacy (perceived confidence) in one's ability to engage in weight control behaviors (e.g., dietary restraint, physical activity) over the next six months will be assessed. Self-efficacy for dietary restraint will be assessed with the short form of the Weight Efficacy Lifestyle Questionnaire (e.g., I can resist eating … when I am depressed or down; 8 items). Self-efficacy for physical activity will be assessed with the Exercise Self-efficacy Scale (e.g., I am confident I can participate in regular exercise when … I am tired; 5 items). Weight control items will be interspersed with items assessing self-efficacy for other health behaviors (e.g., flu vaccination, sleep). Each item will be rated on an 8-point scale (0=not at all confident to 7=very confident). Items will be averaged to create a composite score. Scores will range from 0 to 7, with higher scores indicating higher self-efficacy for weight control behavior.
Time Frame: 6 minutes after delivery of the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Weight Discrimination Experience | Control Experience
Number analyzed (Participants) | 136 | 135
score on a scale | 4.29 (1.42) | 3.91 (1.42)
Statistical Analysis 1: Comparison: Control Experience; Test type: Superiority; p = .029, t-test, 2 sided

4. Primary Outcome: Intentions for Weight Control Behavior
Description: Using the same health behaviors assessed for self-efficacy, intentions for weight control behavior will be assessed (i.e., intentions to engage in each behavior over the next six months). Each item will be rated on an 8-point scale (0=strongly disagree to 7=strongly agree). Items will be averaged to create a composite score. Scores will range from 0 to 7, with higher scores indicating higher intentions to engage in weight control behavior.
Time Frame: 10 minutes after delivery of the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Weight Discrimination Experience | Control Experience
Number analyzed (Participants) | 136 | 135
score on a scale | 4.91 (1.30) | 4.70 (1.28)
Statistical Analysis 1: Comparison: Control Experience; Test type: Superiority; p = .163, t-test, 2 sided

5. Primary Outcome: Executive control_accuracy
Description: The Stroop task provides a measure of executive control by assessing the ability to inhibit an automatic response (reading) in favor of performing a more controlled task (color naming). The task is a classic, widely used and well-validated measure of executive control. Eight blocks of 20 trials will be performed that will take approximately 5 minutes to complete. Executive control scores will be calculated for response accuracy and speed. Metric: accuracy (percentage of correct answers on mismatched trials). A lower percentage of correct answers on mismatched trials indicates worse executive control.
Time Frame: 15 minutes after delivery of the intervention
Population: There are some missing data on this variable due to experimenter error.
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | Weight Discrimination Experience | Control Experience
Number analyzed (Participants) | 132 | 131
percentage of correct responses | 96 (5.0) | 96 (4.7)
Statistical Analysis 1: Comparison: Control Experience; Test type: Superiority; p = .442, t-test, 2 sided

6. Primary Outcome: Executive control_speed
Description: The Stroop task provides a measure of executive control by assessing the ability to inhibit an automatic response (reading) in favor of performing a more controlled task (color naming). The task is a classic, widely used and well-validated measure of executive control. Eight blocks of 20 trials will be performed that will take approximately 5 minutes to complete. Executive control scores will be calculated for accuracy and speed (reaction time). Metric: reaction time (average reaction time in milliseconds on mismatched trials). Longer reaction times on mismatched trials indicate worse executive control.
Time Frame: 15 minutes after delivery of the intervention
Population: There are some missing data on this variable due to experimenter error.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Weight Discrimination Experience | Control Experience
Number analyzed (Participants) | 129 | 133
milliseconds | 1191 (429) | 1362 (492)

7. Primary Outcome: Delay Discounting
Description: Delay discounting involves the subjective depreciation of an incentive based on its timing. The measure assesses the ability to delay gratification, that is, a tendency to prioritize larger long-term rewards over smaller short-term rewards. The task involves choosing short vs. long-term rewards from a set of five dichotomous choices (e.g., to receive $1 immediately or $10 in one month). The task takes about 1 minute to administer, is highly reliable, and correlates well with longer and more extensive measures of delay discounting (metric: discount rate (k)). Scores will range from 0.000110 to 24, with higher scores indicating more impulsivity/lower ability to delay gratification.
Time Frame: 20 minutes after delivery of the intervention
Population: There are some missing data on this variable due to experimenter error.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Weight Discrimination Experience | Control Experience
Number analyzed (Participants) | 133 | 133
score on a scale | 0.86 (3.87) | 1.20 (4.78)
Statistical Analysis 1: Comparison: Control Experience; Test type: Superiority; p = .527, t-test, 2 sided

8. Primary Outcome: Change in Cortisol From Baseline to First Follow-up Assessment
Description: The investigators will measure cortisol secretion via saliva (passive drool) 25 minutes after delivery of the intervention (first follow-up) and compare it to baseline cortisol levels.
Time Frame: 25 minutes after delivery of the intervention
Population: There are some missing data on this variable due to poor quality saliva samples (too watery).
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | Weight Discrimination Experience | Control Experience
Number analyzed (Participants) | 135 | 131
ug/dL | .0000 (.0000) | .0076 (.0874)
Statistical Analysis 1: Comparison: Control Experience; Test type: Superiority; p = .311, t-test, 2 sided

9. Primary Outcome: Comfort Eating
Description: Comfort eating will be assessed via an eating task to objectively measure hyper-palatable (high-fat, -sodium, -sugar, and -carbohydrate) food intake. To avoid floor effects, the eating task will take place under the guise of a faux taste test, which will ostensibly guide the development of the food marketing campaign later during the study. To avoid ceiling effects and to allow eating behavior without fear that the experimenter will negatively judge the amount eaten, large quantities of each food will be made available. The task will take 10 minutes to complete and will be conducted in a private room. Bowls will be weighed (unobtrusively) before and after the task to compute the difference in grams, which will then be converted to kilocalories based on published nutrition information from the food maker. Higher kilocalorie consumption indicates a tendency to engage in more comfort eating during times of stress.
Time Frame: 30 minutes after delivery of the intervention
Population: There are some missing data on this variable due to participant eating restrictions or allergies that prevented them completing the taste test as designed.
Measure: Mean (Standard Deviation); unit: kcals
Arm/Group | Weight Discrimination Experience | Control Experience
Number analyzed (Participants) | 130 | 127
kcals | 299.42 (194.72) | 365.73 (173.83)
Statistical Analysis 1: Comparison: Control Experience; Test type: Superiority; p = .004, t-test, 2 sided

10. Primary Outcome: Social Withdrawal
Description: Social withdrawal will be assessed with a measure from previous research. The experimenter will present three options for working on the final task: alone, with a former group member, or with a new partner. Choosing to work alone reflects a desire to avoid social interaction. Each response will be assigned a numerical code (work alone = 0; work with a former group member = 1; work with a new partner = 2). Scores of zero indicate a greater tendency to withdraw socially during times of stress.
Time Frame: 45 minutes after delivery of the intervention
Population: One participant is missing data due to experimenter error.
Measure: Count of Participants; unit: Participants
Arm/Group | Weight Discrimination Experience | Control Experience
Number analyzed (Participants) | 136 | 134
Participants
  Work by self | 72 | 55
  Work with former group member | 28 | 52
  Work with new group member | 36 | 27
Statistical Analysis 1: Comparison: Control Experience; Test type: Superiority; p = .005, Chi-squared

11. Primary Outcome: Change in Cortisol From Baseline to Second Follow-up Assessment
Description: The investigators will measure cortisol secretion via saliva (passive drool) 60 minutes after delivery of the intervention (second follow-up) and compare it to baseline cortisol levels.
Time Frame: 60 minutes after delivery of the intervention
Population: There are some missing data on this variable due to poor quality saliva samples (too watery). Of note, we were not able to run the statistical analysis on this variable due to the lack of variability in both groups.
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | Weight Discrimination Experience | Control Experience
Number analyzed (Participants) | 135 | 131
ug/dL | .0000 (.0000) | .0000 (.0000)

ADVERSE EVENTS:
Time Frame: 2 hours
Arm/Group | Weight Discrimination Experience | Control Experience
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/135
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/135
Other Adverse Events (participants affected / at risk) | 0/136 | 0/135

LIMITATIONS AND CAVEATS:
Because the of mechanism used to fund this project (R56), we received only one year of funding and thus we were not able to reach our desired sample size of 320 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/96/NCT05714696/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/96/NCT05714696/ICF_001.pdf